CLINICAL TRIAL: NCT01943955
Title: Home-based Computer Gaming in Vestibular Rehabilitation: Effects on Gaze and Balance Impairment
Brief Title: Home-based Computer Gaming in Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS14167
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Peripheral Vestibular Disorders; Vestibular Syndromes &/or Disorders (Labyrinthine); Vestibular Neuronitis
Keywords: dizziness; vertigo; unsteadiness; unbalance; falls
MeSH Terms: conditions — Vestibular Neuronitis; Dizziness; Vertigo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- home-based computer gaming (Experimental): computer gaming, balance exercises carried out at home for 20 minutes 5 days/week and monitored by a physical therapist.
  Interventions: Behavioral: home-based computer gaming

INTERVENTIONS:
Behavioral: home-based computer gaming — A computer mouse mounted to a headband and placed on the participant's head is used to interact with the game cursor. In order to interact with/play the game the participant must visually focus on the moving target and perform unpredictable head movements. Balance exercises are incorporated progressively and simultaneously during computer gaming.
  Other Names: home-based computer gaming for people with PVD

SUMMARY:
It is hypothesized that a home-based computer gaming rehabilitation program will improve gaze control and balance impairments in those with peripheral vestibular disorders (PVD). Ten people with peripheral vestibular disorders were started on a treatment program that consisted of playing computer games and while performing various balance exercises. On a weekly basis, each participant was contacted by email or telephone and asked to submit their computer gaming data to a trained vestibular physical therapist. Following review of this data, the physical therapist would contact the participant and progress their computer gaming program appropriately. At the completion of twelve weeks of home treatment, the participants returned for re-assessment and it was determined that the computer gaming program was an effective treatment for those with PVD. It was also determined that a monitored telerehabilitation program was an efficient and effective delivery method for this treatment.

DETAILED DESCRIPTION:
A pre to post intervention case series study was carried out on ten participants diagnosed with peripheral vestibular disorders (PVD). Inclusion criteria consisted of: a) 20 to 70 year old, b) confirmed diagnosis of PVD on neuro-opthalmic, neuro-orthoptic, electronystagmography and caloric testing; and use of a home computer. Exclusion criteria consisted of those with migraine, central nervous system disorders (for example cerebral vascular accident or Multiple Sclerosis), recent fractures of the spine or lower extremities, inability to stand for 20 minutes continuously, or presence of dementia. It was hypothesized that a home-based computer gaming treatment delivered in a monitored telerehabilitation platform would be an effective treatment for those with PVD in that increased gaze stability and improved balance would be observed post-treatment. It was also hypothesized that decreased dizziness would be reported post-treatment. After initial assessment (pre-treatment), three in-clinic sessions were given to each participant to develop their specific home treatment computer program and ensure ability to use the program effectively. They were then started on their home program and monitored by a trained vestibular physical therapist for a 12-week telerehabilitation program. After the completion of the 12-weeks, the participants returned for a post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of peripheral vestibular disorder (confirmed on electronystagmography, bithermal caloric testing, neuro-ophthalmic, neuro-orthoptic examination)
* Access to a home computer

Exclusion Criteria:

* Central Nervous System disorders
* Vestibular migraine
* Benign Paroxysmal Positional Vertigo (BPPV)
* Recent fractures of the spine or lower extremities
* Inability to tolerate standing for 20 minutes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Centre of Foot Pressure (COP) - Group mean and standard error mean (SEM) of Total Path Length (TPL) in Medial-Lateral and Anterior-Posterior Directions. | Change from baseline in COP at 12 weeks

SECONDARY OUTCOMES:
Trunk Stability - p-value and effect size of trunk root mean square (RMS) angular velocity in Medial-Lateral and Anterior-Posterior directions. | Change from baseline in trunk stability at 12 weeks

OTHER OUTCOMES:
Gaze Stability - group mean and standard error mean (SEM) of open loop (OL) and closed loop (CL) visual tracking tasks during standing on fixed and sponge surfaces and during treadmill walking at 0.7 mph. | change from baseline in gaze stability at 12 weeks
Dizziness - percentiles and p-values for Dizziness Handicap Inventory (DHI) | change from baseline in dizziness at 12 weeks
Gait Stability - percentiles and p-values for Dynamic Gait Index (DGI) | change from baseline in gait stability at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, PhD, Principal Investigator — University of Manitoba; Karen M Reimer, MSc, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, School of Medical Rehabilitation, Winnipeg, Manitoba, Canada